CLINICAL TRIAL: NCT05084469
Title: Exploration of the 5-HT1A Receptor in Cluster Headache : a PET-MRI Study Using the PET Radiopharmaceutical [18F]F13640
Brief Title: Exploration of Cluster Headache in a PET-MRI Study
Acronym: F13640-AVF
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Hospices Civils de Lyon (Other)
Responsible Party: Sponsor
Other Study IDs: 69HCL20_1158; 2021-000209-25 (EudraCT Number)
Record Dates: First submitted 2021-06-09; First posted 2021-10-19 (Actual); Last update posted 2021-10-19 (Actual); Status verified 2021-06

CONDITIONS: Cluster Headache, Episodic
Keywords: Cluster Headache; PET-MRI; 5HT1A
MeSH Terms: conditions — Cluster Headache

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Episodic Cluster Headache patients: Patients will perform two PET-MRI scans: (1) during cluster period and (2) during pain-free remission period. Scans during cluster periods will aim to acquire data before, during and after crisis. Sumatriptan 6mg will be injected subcutaneously under PET-MRI camera to relieve patient pain.
  Interventions: Procedure: PET-MRI in pain-free remission period

INTERVENTIONS:
Procedure: PET-MRI in pain-free remission period — Patients will performed PET-MRI scans. A first 30 minutes acquisition will be performed at time=60min after injection. A second 75 minutes acquisition will be performed at time=150min. Each scans will contain functional dynamic [18F]F13640 PET acquisition, anatomical and functional MRI images acquisition and pain evaluation using a score visual analogic scale.

SUMMARY:
Observational study in PET-MRI using the 5-HT1A agonist PET radiotracer [18F]F13640.

ELIGIBILITY:
Inclusion Criteria:

* Male
* Age between 20 to 45 years old
* Weight between 50 to 90 kg
* No psychiatric or neurologic pathological history
* No cranial trauma history with loss of consciousness
* No juridical protection
* Free and informed consent
* Affiliated with a social security scheme or similar

Exclusion Criteria:

* Subject with present or past dependence on alcohol or any other addictive substance according to the DSM-IV-TR criteria, with the exception of nicotine, caffeine and cannabis
* Subject already participating in another biomedical research project or having participated for less than a year in a study using ionizing radiation
* Subject with a contraindication to MRI exams
* Subject with a contraindication to PET scans using [18F] F13640: hypersensitivity to the active substance or to one of the excipients (sodium chloride)
* Subject with a contraindication to sumatriptan
* Patients with an active infectious disease or associated serious and progressive medical pathology
* Subjects with an inability to understand or carry out the study (language barrier, obvious lack of motivation, etc...) as judged by the investigator
* Patient having exceeded the annual amount of compensation authorized for participation in research protocols.

Ages: 20 Years to 45 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult
Study Population: Male patients with cluster headache episodic and between 20 and 45 years old.
Sampling Method: Non-Probability Sample
Enrollment: 12 (Estimated)
Dates: Start 2021-11-01 (Estimated); Primary Completion 2024-02-01 (Estimated); Study Completion 2024-02-01 (Estimated)

PRIMARY OUTCOMES:
[18F]F13640 binding | 30 minutes From t=60 to t=90 after [18F]F13640 injection on each scans
  Comparison of 5-HT1A density by measuring non-displaceable binding

SECONDARY OUTCOMES:
[18F]F13640 binding | 75 minutes from t=150 to t=225 after [18F]F13640 injection on each scans
  Comparison of 5-HT1A density by measuring non-displaceable binding
MRI images - fMRI | 30 minutes Ffrom t=60 to t=90 a after [18F]F13640 injection on each scans
  Comparison of cerebral activity (fMRI)
MRI images - fMRI | 75 minutes from t=150 to t=225 after [18F]F13640 injection on each scans
  Comparison of cerebral activity (fMRI)
MRI images - perfusion MRI | 30 minutes from t=60 to t=90 after [18F]F13640 injection on each scans
  Comparison of cerebral blood flow (perfusion MRI).
MRI images - perfusion MRI | 75 minutes from t=150 to t=225 after [18F]F13640 injection on each scans
  Comparison of cerebral blood flow (perfusion MRI).
MRI images - BOLD signal | 30 minutes from t=60 to t=90 after [18F]F13640 injection on each scans
  Comparison of functional connectivity (BOLD signal).
MRI images - BOLD signal | 75 minutes from t=150 to t=225 after [18F]F13640 injection on each scans
  Comparison of functional connectivity (BOLD signal).
Change in general anxiety | baseline
  Hospital Anxiety and Depression scale. Scores range from 0 to 21. Scores with 7 or less are considered as normal. Scores 8 to 10 as borderline abnormal and 11 to 21 as abnormal (case).
Change in general anxiety | day of imaging visit at pain-free remission period up to 24 months after inclusion
  Hospital Anxiety and Depression scale. Scores range from 0 to 21. Scores with 7 or less are considered as normal. Scores 8 to 10 as borderline abnormal and 11 to 21 as abnormal (case).
Change in general anxiety | day of imaging visit during cluster period up to 24 months after inclusion
  Hospital Anxiety and Depression scale. Scores range from 0 to 21. Scores with 7 or less are considered as normal. Scores 8 to 10 as borderline abnormal and 11 to 21 as abnormal (case).
Mood changing (depression) | baseline
  Hospital Anxiety and Depression scale. Scores range from 0 to 21. Scores with 7 or less are considered as normal. Scores 8 to 10 as borderline abnormal and 11 to 21 as abnormal (case).
Mood changing (depression) | day of imaging visit at pain-free remission period up to 24 months after inclusion
  Hospital Anxiety and Depression scale. Scores range from 0 to 21. Scores with 7 or less are considered as normal. Scores 8 to 10 as borderline abnormal and 11 to 21 as abnormal (case).
Mood changing (depression) | day of imaging visit during cluster period up to 24 months after inclusion.
  Hospital Anxiety and Depression scale. Scores range from 0 to 21. Scores with 7 or less are considered as normal. Scores 8 to 10 as borderline abnormal and 11 to 21 as abnormal (case).
Evaluation of pain | During PET-MRI scans, 30 minutes from t=60 to t=90 after [18F]F13640 injection
  Evaluation of pain during days of PET-MRI using a VAS projected on a screen in the camera (0= no pain; 10= pain as bad as can be)
Evaluation of pain | During PET-MRI scans, 75 minutes from t=150 to t=225 after [18F]F13640 injection
  Evaluation of pain during days of PET-MRI using a VAS projected on a screen in the camera (0= no pain; 10= pain as bad as can be)
Acute anxiety | At five points during the day : (1) before scans, (2) time =70minutes, (3) time =105minutes, (4) time=155 minutes, (5) time=240 minutes
  Evaluation of acute anxiety during days of PET-MRI using a VAS questionnaire (0= no anxiety; 10= anxiety as bad as can be)

CONTACTS AND LOCATIONS:
Overall Officials: Genevieve Demarquay, MD, Principal Investigator — Centre d'évaluation et traitement de la douleur